CLINICAL TRIAL: NCT06016413
Title: A Prospective, Single-arm, Phase II Study of Adelbelimab Combined With Carboplatin and Nab-paclitaxel in Neoadjuvant Therapy for Patients With Resectable Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Adelbelimab Combination Chemotherapy in Neoadjuvant Therapy for Squamous Cell Carcinoma of the Head and Neck
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-616-02
Record Dates: First submitted 2023-08-07; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: head and neck squamous cell carcinoma; immunity therapy; PD-L1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Taxes; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): All patients received nab-paclitaxel 260 mg/m2, carboplatin AUC=5 and adelbelimumab 1200 mg intravenously on day 1 of each 3-week cycle for 3 cycles. All patients were given conventional drugs to prevent vomiting in each cycle, and intravenous dexamethasone was given to prevent allergy before each dose
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin; Drug: adelbelimumab

INTERVENTIONS:
Drug: Nab paclitaxel — All patients received nab-paclitaxel 260 mg/m2 intravenously on day 1 of each 3-week cycle for 3 cycles.
Drug: Carboplatin — All patients received carboplatin AUC=5 intravenously on day 1 of each 3-week cycle for 3 cycles.
Drug: adelbelimumab — All patients received carboplatin AUC=5 intravenously on day 1 of each 3-week cycle for 3 cycles.

SUMMARY:
This study explored the efficacy of adelbelimab (PD-L1 inhibitor) combined with chemotherapy in preoperative induction chemotherapy in patients with locally advanced head and neck squamous cell carcinoma

DETAILED DESCRIPTION:
According to the latest data from the International Agency for Research on Cancer, the new incidence of head and neck cancer in the world in 2022 will be among the top ten new incidences of cancer in the world. In the latest WHO classification of head and neck tumors, head and neck cancers include nasopharyngeal cancer, oral cavity cancer, oropharyngeal cancer, thyroid cancer, laryngeal cancer and other malignant tumors that occur in the head and neck, of which more than 90% are squamous cells cancer. Currently, the standard of care for locally advanced head and neck squamous cell carcinoma (HNSCC) is surgical resection followed by risk-adapted adjuvant radiotherapy, with or without platinum-based chemotherapy, or definitive concurrent chemoradiotherapy. With this aggressive combination therapy, the risk of recurrence, distant metastasis, and death remains high in patients with locally advanced human papillomavirus (HPV)-negative HNSCC. In terms of preoperative induction chemotherapy, clinical studies have shown that patients with tumor remission after preoperative induction chemotherapy have a higher survival rate and a lower risk of distant metastasis, but the postoperative pathological complete remission rate of the tumor is lower , it is difficult to be satisfactory. With the rise of tumor immunology, more and more immunotherapy methods are applied to the clinical treatment of tumors. Current immunotherapies come in many forms, including immune checkpoint inhibitors, co-stimulatory point agonists, antigen vaccines, oncolytic virus therapy, adoptive T cell transfer (ACT) and epidermal growth factor receptor ( Epidermal growth factor receptor, EGFR) targeted therapy. Among them, immune checkpoint inhibitors have been widely used in the clinical treatment of tumors, and the molecular mechanisms of immune checkpoints (immune checkpoint inhibitors, ICIs) are mainly such as programmed cell death 1 (PD-1) and cytotoxic T lymphocytes. Cellular antigen 4 (CTLA-4) is a co-inhibitory receptor expressed on the surface of T cells to negatively regulate T cell-mediated immune responses; however, tumor cells utilize these inhibitory molecules to induce tumor tolerance and T cell exhaustion. Therefore, ICIs such as anti-CTLA-4, anti-PD-1, and anti-PD-L1 can attach to these co-inhibitory receptors to reactivate the immune response against tumor cells. In head and neck squamous cell carcinoma, immune checkpoint inhibitors have been widely used clinically, among which PD-1 inhibitors are the most widely used. A clinical study (KEYNOTE-048) showed that pembrolizumab combined with chemotherapy can significantly improve the survival time of recurrent and metastatic head and neck squamous cell carcinoma. And this is also included in the first-line recommendation of the NCCN guidelines for the treatment of patients with recurrent and metastatic head and neck squamous cell carcinoma. In terms of preoperative neoadjuvant chemotherapy for head and neck squamous cell carcinoma, camrelizumab combined with chemotherapy neoadjuvant chemotherapy in the treatment of locally advanced HNSCC showed high objective response rate and pathological response rate. PD-L1 and PD-L2 are two ligands of PD-1. Both tumor and immune cells can express PD-L1, and PD-L1 is a useful biomarker to predict the response to PD-1/PD-L1 antibodies in patients with different types of cancer. PD-L1 plays a role in inhibiting the cancer-immune cycle by binding to negative regulators of T cell activation such as PD-1 and B7.1. However, PD-L1 inhibitors are currently less used in clinical tumor treatment, mainly focusing on small cell lung cancer. Among them, adelbelimab is a human monoclonal antibody against programmed death ligand 1 (PD-L1), and its safety has been verified to some extent. In a multicenter, randomized, double-blind, placebo-controlled phase 3 clinical trial, the median follow-up time of the test group was 13.5 months and the placebo group was 12.8 months; the hazard ratio was 0.72 [95% confidence interval 0.58-0.90]; Compared with one-sided p=0.017), the median overall survival rate of the adelbelimab group was significantly improved (median 15.3 months [95% CI 13.2-17.5]) . In terms of head and neck squamous cell carcinoma, only phase I clinical studies have confirmed the safety and tumor activity of PD-L1 inhibitors in treatment. On this basis, this study will further verify the efficacy of preoperative neoadjuvant chemotherapy in patients with resectable locally advanced head and neck squamous cell carcinoma with PD-L1 inhibitors combined with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-75 years old
2. According to the 8th edition of the guidelines of the American Joint Committee on Cancer (AJCC), patients with stage III-IVB tumors of non-oropharyngeal cancers confirmed by pathology as head and neck squamous cell carcinoma (oral cavity, oropharynx, hypopharynx or larynx) and HPV-negative oropharyngeal cancer patients, or HPV-positive oropharyngeal cancer patients with stage II-III tumors
3. Resectable tumors were evaluated by head and neck surgeons before enrollment to exclude clinical evidence of distant metastasis
4. According to RECIST 1.1, there is at least one measurable tumor lesion
5. The performance status of the Eastern Cooperative Oncology Group (ECOG) is 0-1
6. Blood routine: white blood cell count (WBC) ≥ 3.0×109/L; absolute neutrophil count (ANC) ≥ 1.5×109/L; platelet (PLT) ≥ 100×109/L; hemoglobin level (HGB) ≥ 9.0 g/dL (without corresponding supportive treatment such as blood transfusion and leukocytosis within 7 days).
7. Liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) in patients without liver metastasis ≤ 2.5 times the upper limit of the reference value (ULN); albumin (ALB) ≥ 30 g /L.
8. Renal function: serum creatinine ≤ 1.5 times ULN or creatinine clearance (CrCl) ≥ 50mL/min (using the Cockcroft/Galter formula); urine protein (UPRO) < (++), or 24 Hourly urine protein < 1.0 g.
9. Determination of HPV status in oropharyngeal cancers using p16 IHC. A sample was considered p16 positive if >70% of tumor cells exhibited intense diffuse nuclear and cytoplasmic staining
10. Have not participated in other clinical trial projects in the past 30 days;
11. Patients who voluntarily participate in the project and sign the informed consent.

Exclusion Criteria:

1. The patient has abnormal blood indicators, abnormal liver and kidney function, and cannot tolerate the clinical research process after multidisciplinary consultation evaluation
2. The patient has previously suffered from other tumors, or has previously undergone anti-tumor treatments such as surgery, chemotherapy, and radiotherapy
3. The entire clinical research process cannot be completed due to personal, social and economic reasons
4. Serious systemic diseases in the past and the diseases cannot be cured or controlled by drugs -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pathological complete response rate | one week after operative
  The postoperative specimens were sent to the pathology department for fixation, sectioning, and observation. Two pathologists judge whether the subject's tumor remains. If there is a disagreement between the two, the third senior pathologist will discuss and decide

SECONDARY OUTCOMES:
Major pathological response rate | one week after operative
  The postoperative specimens were sent to the pathology department for fixation, sectioning, and observation. Two pathologists judge whether the subject's tumor remains. If there is a disagreement between the two, the third senior pathologist will discuss and decide
Two years overall Survival | Two years after investigator enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Colevas AD, Bahleda R, Braiteh F, Balmanoukian A, Brana I, Chau NG, Sarkar I, Molinero L, Grossman W, Kabbinavar F, Fasso M, O'Hear C, Powderly J. Safety and clinical activity of atezolizumab in head and neck cancer: results from a phase I trial. Ann Oncol. 2018 Nov 1;29(11):2247-2253. doi: 10.1093/annonc/mdy411. PMID 30219915
- [Background] Wang J, Zhou C, Yao W, Wang Q, Min X, Chen G, Xu X, Li X, Xu F, Fang Y, Yang R, Yu G, Gong Y, Zhao J, Fan Y, Liu Q, Cao L, Yao Y, Liu Y, Li X, Wu J, He Z, Lu K, Jiang L, Hu C, Zhao W, Zhang B, Shi W, Zhang X, Cheng Y; CAPSTONE-1 Study Group. Adebrelimab or placebo plus carboplatin and etoposide as first-line treatment for extensive-stage small-cell lung cancer (CAPSTONE-1): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2022 Jun;23(6):739-747. doi: 10.1016/S1470-2045(22)00224-8. Epub 2022 May 13. PMID 35576956
- [Background] Herbst RS, Soria JC, Kowanetz M, Fine GD, Hamid O, Gordon MS, Sosman JA, McDermott DF, Powderly JD, Gettinger SN, Kohrt HE, Horn L, Lawrence DP, Rost S, Leabman M, Xiao Y, Mokatrin A, Koeppen H, Hegde PS, Mellman I, Chen DS, Hodi FS. Predictive correlates of response to the anti-PD-L1 antibody MPDL3280A in cancer patients. Nature. 2014 Nov 27;515(7528):563-7. doi: 10.1038/nature14011. PMID 25428504
- [Background] Doroshow DB, Bhalla S, Beasley MB, Sholl LM, Kerr KM, Gnjatic S, Wistuba II, Rimm DL, Tsao MS, Hirsch FR. PD-L1 as a biomarker of response to immune-checkpoint inhibitors. Nat Rev Clin Oncol. 2021 Jun;18(6):345-362. doi: 10.1038/s41571-021-00473-5. Epub 2021 Feb 12. PMID 33580222
- [Background] Wu Y, Chen W, Xu ZP, Gu W. PD-L1 Distribution and Perspective for Cancer Immunotherapy-Blockade, Knockdown, or Inhibition. Front Immunol. 2019 Aug 27;10:2022. doi: 10.3389/fimmu.2019.02022. eCollection 2019. PMID 31507611
- [Background] Zhang Z, Wu B, Peng G, Xiao G, Huang J, Ding Q, Yang C, Xiong X, Ma H, Shi L, Yang J, Hong X, Wei J, Qin Y, Wan C, Zhong Y, Zhou Y, Zhao X, Leng Y, Zhang T, Wu G, Yao M, Zhang X, Yang K. Neoadjuvant Chemoimmunotherapy for the Treatment of Locally Advanced Head and Neck Squamous Cell Carcinoma: A Single-Arm Phase 2 Clinical Trial. Clin Cancer Res. 2022 Aug 2;28(15):3268-3276. doi: 10.1158/1078-0432.CCR-22-0666. PMID 35766967
- [Background] Burtness B, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Hong RL, Gonzalez Mendoza R, Roy A, Zhang Y, Gumuscu B, Cheng JD, Jin F, Rischin D; KEYNOTE-048 Investigators. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019 Nov 23;394(10212):1915-1928. doi: 10.1016/S0140-6736(19)32591-7. Epub 2019 Nov 1. PMID 31679945
- [Background] Seidel JA, Otsuka A, Kabashima K. Anti-PD-1 and Anti-CTLA-4 Therapies in Cancer: Mechanisms of Action, Efficacy, and Limitations. Front Oncol. 2018 Mar 28;8:86. doi: 10.3389/fonc.2018.00086. eCollection 2018. PMID 29644214
- [Background] Sadeghi Rad H, Monkman J, Warkiani ME, Ladwa R, O'Byrne K, Rezaei N, Kulasinghe A. Understanding the tumor microenvironment for effective immunotherapy. Med Res Rev. 2021 May;41(3):1474-1498. doi: 10.1002/med.21765. Epub 2020 Dec 4. PMID 33277742
- [Background] Yu C, Li Q, Zhang Y, Wen ZF, Dong H, Mou Y. Current status and perspective of tumor immunotherapy for head and neck squamous cell carcinoma. Front Cell Dev Biol. 2022 Aug 26;10:941750. doi: 10.3389/fcell.2022.941750. eCollection 2022. PMID 36092724
- [Background] Zhong LP, Zhang CP, Ren GX, Guo W, William WN Jr, Sun J, Zhu HG, Tu WY, Li J, Cai YL, Wang LZ, Fan XD, Wang ZH, Hu YJ, Ji T, Yang WJ, Ye WM, Li J, He Y, Wang YA, Xu LQ, Wang BS, Kies MS, Lee JJ, Myers JN, Zhang ZY. Randomized phase III trial of induction chemotherapy with docetaxel, cisplatin, and fluorouracil followed by surgery versus up-front surgery in locally advanced resectable oral squamous cell carcinoma. J Clin Oncol. 2013 Feb 20;31(6):744-51. doi: 10.1200/JCO.2012.43.8820. Epub 2012 Nov 5. PMID 23129742
- [Background] Bernier J, Domenge C, Ozsahin M, Matuszewska K, Lefebvre JL, Greiner RH, Giralt J, Maingon P, Rolland F, Bolla M, Cognetti F, Bourhis J, Kirkpatrick A, van Glabbeke M; European Organization for Research and Treatment of Cancer Trial 22931. Postoperative irradiation with or without concomitant chemotherapy for locally advanced head and neck cancer. N Engl J Med. 2004 May 6;350(19):1945-52. doi: 10.1056/NEJMoa032641. PMID 15128894
- [Background] Cooper JS, Pajak TF, Forastiere AA, Jacobs J, Campbell BH, Saxman SB, Kish JA, Kim HE, Cmelak AJ, Rotman M, Machtay M, Ensley JF, Chao KS, Schultz CJ, Lee N, Fu KK; Radiation Therapy Oncology Group 9501/Intergroup. Postoperative concurrent radiotherapy and chemotherapy for high-risk squamous-cell carcinoma of the head and neck. N Engl J Med. 2004 May 6;350(19):1937-44. doi: 10.1056/NEJMoa032646. PMID 15128893
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204